CLINICAL TRIAL: NCT06560866
Title: Disrupting Social Risk Factors of Health to Improve Substance Use and Mental Health Outcomes for Parents in Rural Regions
Brief Title: Disrupting SRFOH to Improve Substance Use and Mental Health Outcomes for Parents in Rural Regions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lisa Saldana, Research Scientist, Chestnut Health Systems
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1172-0623; R01DA057556 (NIH)
Record Dates: First submitted 2024-07-10; First posted 2024-08-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-08

CONDITIONS: Substance-Related Disorders
Keywords: social risk factors; opioid; methamphetamine; child welfare; prevention; evidence-based
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: This study is a single group intensive longitudinal observational study. This is not a randomized trial. All participants will receive Just Care for Families treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Just Care for Families (Experimental): Parents receiving Just Care for Families
  Interventions: Behavioral: Just Care for Families

INTERVENTIONS:
Behavioral: Just Care for Families — Just Care for Families is a behavioral intervention to address the needs of families involved in or at-risk for involvement with the child welfare system. Just Care involves treatment components, supported by ongoing purposeful engagement: (1) Substance use treatment including contingency management and positive reinforcement, day planning, healthy environments and peer choices, and refusal skills; (2) Mental health treatment including cognitive behavioral therapy, developing healthy coping skills, emotion regulation skills, exposure therapy, and referral for medication management; (3) Parent management training including parenting skills, nurturing and attachment, reinforcement, emotion regulation, supervision, structure, non-harsh discipline, and nutrition; (4) Community building including indigenous and external social supports; (5) Systems navigation; and (6) provision of assistance with basic needs including assistance with housing and employment.

SUMMARY:
The study will evaluate the effectiveness of the Just Care for Families program in preventing Oregon Department of Human Services (ODHS)-involved parents in rural communities from escalating opioid and/or methamphetamine use and mental health disorders by disrupting the associated social risk factors of health (SRFOH). In addition, investigators will examine the impacts of SRFOH on Just Care treatment and the associated costs from the perspective of provider clinics delivering Just Care. Just Care is a behavioral intervention for the treatment of parental substance abuse and child neglect for families involved in the child welfare system. Just Care involves treatment components, supported by ongoing purposeful engagement: (1) Substance use treatment; (2) Mental health treatment; (3) Parent management training; (4) Community building; (5) Systems Navigation; and (6) Addressing basic needs.

DETAILED DESCRIPTION:
This study provides multiple tests of the mechanisms by which Just Care for Families disrupts the effects of lifetime social risk factors of health (SRFOH) on ultimate outcomes of preventing escalation of opioid and/or methamphetamine use and suicide (ideation, intention, attempts). Just Care for Families 's effect on these outcomes is hypothesized to occur through two mechanisms of action: (1) improvement in malleable SRFOH (direct targets of intervention) and (2) improvement in substance use and mental health problems (intermediate prevention outcomes). Analyses will examine whether the effects vary as a function of non-malleable external, structural SRFOH, such as community poverty and healthcare service availability. Additionally, system dynamics will be used to examine patterns of influence between SRFOH and Just Care for Families intervention targets, case outcomes, and associated costs.

ELIGIBILITY:
Inclusion Criteria:

Parents:

* Any substance misuse in the last year
* Parent of a child, age 0-18
* Resident of participating county (Lane, Linn, Benton, Douglas, Lincoln)
* Insured by Oregon Health Plan (Medicaid)
* Access to a computer or smartphone; or wireless/cellular connection if a device were to be provided; or reliable access to a landline to receive a brief weekly phone assessment in place of the digital assessment

Clinical Staff:

* clinician at a participating clinic
* Providing Just Care for Families services to parents in the study at any point during study

Exclusion Criteria:

* Alcohol use disorder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in opioid use | baseline, 9 months, and 18 months
  Changes in any opioid use in past 30 days as assessed by Addiction Severity Index opioid use items (heroin, methadone, and other).
Change in methamphetamine use | baseline, 9 months, 18 months
  Changes in any methamphetamine use in past 30 days as assessed by Addiction Severity Index.
Change in depression severity | Baseline, 9 months and 18 months
  Changes in intensity of depression-related distress in the past week as measured by the Brief Symptom Inventory Depression Subscale items (Sum of responses to 6 Likert-type items, range 0-24).
Change in anxiety | baseline, 9 months, 18 months
  Changes in intensity of anxiety-related distress in the past week as measured by the Brief Symptom Inventory Anxiety Subscale items (Sum of responses to 6 Likert-type items, range 0-24).
Change in Social Risk Factors Needs | Baseline through 18 months (weekly)
  Changes in total number of needs or problems across Social Risk Factors of Health domains as assessed by PhenX toolkit items in a weekly parent survey. The number of items endorsed in the past week out of 43 items comprising 7 risk factor domains are scored. Domains include Work and money, neighborhood and transportation, education and training, food, community safety and support, healthcare system, internet and phone, and health and well-being.

SECONDARY OUTCOMES:
Changes in opioid or methamphetamine use as measured by Urinalysis testing | Baseline through 18 months (weekly)
  Positive urine drug screen for opioids or methamphetamines as measured by 12-panel instant urine toxicology screens and fentanyl strip screens.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Saldana, PhD, Principal Investigator — Chestnut Health Systems
Locations (1):
- Chestnut Health Systems, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
As part of the NIH Helping to End Addiction Long-term (HEAL) Initiative, this study will follow the data sharing protocols as outlined by the HEAL Data Sharing Policy.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be shared upon acceptance of the data for publication or within six months after the completion of Baseline data collection (within 12 months for the 9-month and 18-month assessments), whichever is earlier.
Access Criteria: Data will be deposited in the NAHDAP data repository. These data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and could be used for secondary study purposes. Requested primary study data and metadata will be made available to investigators according to the policies of the NAHDAP.

DOCUMENTS (1):
  • Informed Consent Form (2024-10-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT06560866/ICF_001.pdf